CLINICAL TRIAL: NCT00510692
Title: A Two-Arm Chemoprevention Trial in Familial Adenomatous Polyposis (FAP) Coli Patients Using the Purified Free Fatty Acid, Eicosapentaenoic Acid
Brief Title: Chemoprevention Trial in Familial Adenomatous Polyposis (FAP) Coli Using EPA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: S.L.A. Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EPA/POL/03
Record Dates: First submitted 2007-07-30; First posted 2007-08-02 (Estimated); Results first posted 2014-08-22 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Familial Adenomatous Polyposis Coli; FAP
Keywords: Eicosapentaenoic Acid; EPA; EPA 99%; Fatty acid; omega-3; apoptosis; cell proliferation; colonic mucosa; polyp; Familial Adenomatous Polyposis Coli; FAP; resolvin; Ileo-rectal anastomosis; IRA; PUFA; Endoscopy
MeSH Terms: conditions — Adenomatous Polyposis Coli; Hyperplasia; Polyps | interventions — Eicosapentaenoic Acid; Endoscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2g/day Eicosapentanoic Acid (EPA) (Experimental): Eicosapentanenoic Acid (EPA) as the free fatty acid 2 capsules twice daily for 6 months.
  Endoscopy and biopsies taken as described under intervention.
  Interventions: Drug: Eicosapentanoic Acid (EPA); Procedure: Endoscopy; Procedure: Biopsies taken
- Placebo (Placebo Comparator): Medium chain triglycerides 2 capsules twice daily for six months. Endoscopy and biopsies taken as described under intervention.
  Interventions: Procedure: Endoscopy; Procedure: Biopsies taken; Drug: Placebo

INTERVENTIONS:
Drug: Eicosapentanoic Acid (EPA) — 2 x 500mg EPA capsules twice daily for 6 months
  Other Names: ALFA
  Arms: 2g/day Eicosapentanoic Acid (EPA)
Procedure: Endoscopy — Endoscopy with video and photographs at baseline and month 6.
  Other Names: Endoscopy either Colonoscopy or Flexible sigmoidoscopy.
Procedure: Biopsies taken — 9 biopsies taken at baseline and month 6 from the rectum of normal mucosa for analysis of apoptosis (3 biopsies), cell proliferation (3 biopsies) and mucosal fatty acid levels (3 biopsies). Two biopsies taken at baseline and month 6 from polyps for cell proliferation (1 biopsy) and apoptosis (1 biopsy).
Drug: Placebo — 2 x 500mg placebo capsules twice daily for 6 months
  Arms: Placebo

SUMMARY:
This purpose of this study is to investigate whether the number and size of rectal polyps can be reduced in patients with Familial Adenomatous Polyposis (FAP) by using a highly-purified form of a naturally occurring substance, the omega-3 fatty acid, eicosapentaenoic acid (EPA).

DETAILED DESCRIPTION:
It has been found that people who consume a large amount of oily fish tend to have a lower risk of developing colon cancer. This is thought to be due to the omega-3 fatty acids present in oily fish, one of which is EPA. The effect of taking a 99% pure form of EPA (2g per day) compared with placebo capsules on the number and size of polyps in the rectum over a six month period will be investigated.

FAP is an inherited susceptibility to diffuse colorectal adenomas and colorectal carcinoma, occurring in close to 100% of unresected colons. It is caused by a germline mutation in the Adenomatous Polyposis Coli (APC) gene located in the long arm of chromosome 5. To prevent cancer development it is recommended that patients with FAP undergo colectomy with ileo-anal or ileo-rectal anastomosis (or colectomy and end-ileostomy) at a socially convenient time before polyp progression to malignancy and before the age of 25. Patients with the attenuated FAP phenotype, often associated with mutations at the 5' terminus (exon 4 and proximally), have fewer polyps and may often delay colectomy. Patients with an ileo-rectal anastomosis are still susceptible to polyp formation in the remaining rectal stump and require 6 monthly check-ups with a flexible sigmoidoscope with removal of any polyps that develop. Therefore, an effective chemopreventative agent with a favourable side-effect profile would be of benefit to FAP patients with ileo-rectal anastomosis (IRA) and recurrent rectal polyps in addition to young adults who prefer to delay colectomy. If such an agent were to be effective in FAP patients in the prevention of colonic polyps, it may also be of benefit to the larger population of patients with sporadic colorectal adenomatous polyps who are also at risk of colorectal cancer.

Colorectal polyps are thought, at least in part, to arise from an imbalance in the levels of cell proliferation and apoptosis (natural cell death) in the colonic mucosa. It has been suggested that omega-3 polyunsaturated fatty acids (PUFAs) in fish oil can manipulate the high levels of colonic-mucosal cell proliferation rates associated with colonic adenomas.

The rationale for this trial is based on the increasing evidence linking inflammatory processes and the development of a number of cancers, including bowel cancer. This has focused attention on the role of inflammatory mediators in the development of cancer. In particular, the family of eicosanoids (including 2-series prostaglandins, 4-series leukotrienes and thromboxanes) produced through conversion of the omega-6 PUFA, arachidonic acid, via cyclo-oxygenase-2 (COX-2) is believed to contribute to the physiological processes of inflammation and the development of tumours. Prostaglandin E2, a product of the conversion of arachidonic acid via the COX-2 pathway, has been implicated in tumourigenesis through:

1. promotion of angiogenesis
2. anti-apoptotic properties
3. increasing expression of matrix metalloproteinases and hence the ability of a tumour cell to undergo metastasis
4. altering the cytokine expression profile of cells.

The class of eicosanoid synthesised will depend on the PUFA substrate. Whilst arachidonic acid is converted to 2-series prostaglandins and 4-series leukotrienes, EPA is converted to 3-series prostaglandins and 5-series leukotrienes. Overall, the latter eicosanoids are less potent as inflammatory mediators than those derived from arachidonic acid.

Increasing daily intake of EPA, the omega-3 PUFA analogue of arachidonic acid, alters the balance between the cell content of these fatty acids. This results in reduced production of the more active inflammatory/tumourigenic products of arachidonic acid metabolism. This is supported by the results of recent work at St George's Hospital Medical School, London. In patients with a history of colonic adenomas, daily dosing with a highly purified, free-fatty acid form of the EPA produced a significant reduction in cell proliferation and increase in apoptosis in the colonic mucosa. This preparation of EPA has the proprietary name "Alfa" and is referred to here as EPA.

This proposed study will be based upon the randomised, placebo-controlled National Cancer Institute sponsored study in which three groups of FAP patients were assigned to one of two doses of celecoxib (a COX-2 inhibitor) or placebo. The results showed a reduction in the polyp burden of the group taking the higher (400mg twice daily (bd)) dose. However, there is evidence to suggest that COX-2 inhibitors carry significant potential for side-effects. Adopting a similar design, EPA will be substituted for celecoxib in this randomised, placebo-controlled trial, comparing 2g EPA to placebo, with reduction in polyp burden as the primary objective.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a known diagnosis of Familial Adenomatous Polyposis (FAP) and have had a previous colectomy with ileo-rectal anastomosis.
* Males or females aged 18 and over
* If the participant is female and of child bearing potential, she agrees to participate in this study by providing written informed consent, has been using adequate contraception (e.g. abstinence, condom, Intra-uterine device (IUD), birth control pill, diaphragm and spermicidal gel combination) since her last menses and will use adequate contraception during the study, is not lactating, and agrees to undergo a serum pregnancy test at baseline and month 6. Sexually active males must agree to use an accepted method of contraception.
* Rectal polyp status: the subject has an endoscopically assessable rectal segment.
* Subjects must show a willingness to abstain from regular use of non-steroidal anti-inflammatory medication for the duration of the study. A cardioprotective dose of aspirin (75mg) will be permitted.
* Subjects must have provided written informed consent to participate.
* Subjects must have assessable rectal polyps post baseline flexible sigmoidoscopy.
* Subjects must have the following rectal polyp burden at the conclusion of the baseline endoscopy:
* Rectum - 3 or more quantifiable polyps ≥2mm diameter
* In the rectum quantifiable polyps are defined as being within a composite "cloverleaf" photograph that includes a tattoo.

Exclusion Criteria:

* Subjects who are due to undergo an anticipated colectomy within 8 months of randomisation
* History of invasive carcinoma in the past 5 years other than resected Dukes' A/B1 colon cancer or resected non-melanomatous skin cancer
* Partial or complete colectomy within 12 months prior to enrolment.
* History of pelvic radiation
* Subjects who are allergic to fish
* Subjects who have diabetes mellitus
* Subjects who are pregnant or breast-feeding
* Subjects taking aspirin or other non-steroidal anti-inflammatory drugs on a regular basis other than low dose (75 mg) cardioprotective dose.
* Subjects who have aspirin-sensitive asthma
* Subjects suffering from haemorrhagic disorders
* Subjects who are taking warfarin or other anticoagulants
* Subjects who have significant abnormalities on their screening blood tests
* Subjects taking lipid lowering medication
* Subjects with gastrointestinal malabsorptive disease
* Subjects with known or prior coagulopathy
* Subjects with uncontrolled hypercholesterolaemia
* Subjects who are taking other fish-oil supplements (e.g. cod liver oil) who are unwilling to stop them for the duration of the study. Subjects previously taking fish oil must have a washout period of 1 month prior to study enrolment.
* Subjects who are deemed mentally incompetent, or have a history of anorexia nervosa or bulimia
* Subjects with a history of alcohol or drug abuse, including laxative abuse which would render the subject unreliable.
* Subjects considered by their physician unlikely to be able to comply with the protocol.
* Subjects who have taken part in an experimental drug study in the preceding 3 months.
* Subjects who have a positive pregnancy test within 14 days prior to baseline visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2006-11; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas J West, MB BS FRCS, Principal Investigator — The Polyposis Registry, St. Mark's Hospital,
Locations (1):
- The Polyposis Registry, St. Mark's Hospital,, Harrow, Middlesex, United Kingdom

REFERENCES:
- [Derived] West NJ, Clark SK, Phillips RK, Hutchinson JM, Leicester RJ, Belluzzi A, Hull MA. Eicosapentaenoic acid reduces rectal polyp number and size in familial adenomatous polyposis. Gut. 2010 Jul;59(7):918-25. doi: 10.1136/gut.2009.200642. Epub 2010 Mar 26. PMID 20348368

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Single centre study (Polyposis Registry).
Groups:
- 2g/Day Eicosapentaenoic Acid (EPA): Eicosapentaenoic Acid (EPA) 2g per day for six months
- Placebo: Medium chain triglycerides 2 g per day for six months.
Period: Overall Study
Arm/Group | 2g/Day Eicosapentaenoic Acid (EPA) | Placebo
Started | 29 | 29
Completed | 27 | 26
Not Completed | 2 | 3
Not completed — Adverse Event | 1 | 3
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: The baseline characteristics are presented for the full analysis set which constitutes 55 of the 58 randomised subjects. The full analysis set includes all subjects who were randomised into the study, took at least one dose of study medication provided both at baseline and at least one treatment measurement for efficacy.
Groups:
- 2g/Day EPA: Eicosapentanoic Acid (EPA): 2 x 500mg EPA capsules twice daily for 6 months
  Endoscopy: With video and photographs at baseline and month 6.
  Biopsies taken: 9 biopsies taken at baseline and month 6 from the rectum of normal mucosa for analysis of apoptosis (3 biopsies), cell proliferation (3 biopsies) and mucosal fatty acid levels (3 biopsies). Two biopsies taken at baseline and month 6 from polyps for cell proliferation (1 biopsy) and apoptosis (1 biopsy).
- Placebo: Medium chain triglycerides 2 capsules twice daily for six months.
  Endoscopy: With video and photographs at baseline and month 6.
  Biopsies taken: 9 biopsies taken at baseline and month 6 from the rectum of normal mucosa for analysis of apoptosis (3 biopsies), cell proliferation (3 biopsies) and mucosal fatty acid levels (3 biopsies). Two biopsies taken at baseline and month 6 from polyps for cell proliferation (1 biopsy) and apoptosis (1 biopsy).
- Total: Total of all reporting groups
Arm/Group | 2g/Day EPA | Placebo | Total
Number analyzed (Participants) | 28 | 27 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (11.4) | 42.5 (13.8) | 40.1 (12.6)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 26 | 54
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 27
  Male | 13 | 15 | 28
Region of Enrollment [Number; unit: participants]
  United Kingdom | 28 | 27 | 55

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in the Number of Polyps Measured in a Focal Area of the Rectum.
Description: Absolute change in the number of polyps measured in a defined focal area of the rectum.
Time Frame: 6 months compared to baseline.
Population: 13 subjects lacked the photographs required for counting the measurements of polyps. Reasons for lack of photographs varied including failure of video equipment, inability to identify identical views of the focal area and no forceps visible for calibration.
Measure: Mean (Standard Deviation); unit: Change from baseline number of polyps.
Groups:
- Placebo: Medium chain triglycerides 2g per day for six months
Arm/Group | 2g/Day Eicosapentaenoic Acid (EPA) | Placebo
Number analyzed (Participants) | 23 | 22
Change from baseline number of polyps. | -0.5 (0.9) | 0.5 (1.4)
Statistical Analysis 1: Comparison: 2g/Day Eicosapentaenoic Acid (EPA) vs Placebo; Test type: Superiority or Other; p = 0.005, ANCOVA; Mean Difference (Net) = -1.06, 95% CI 2-sided [-1.78 to -0.35]

2. Secondary Outcome: Percentage Change in the Number of Polyps Measured in the Defined Focal Area of the Rectum.
Description: Percentage change in the number of polyps measured in the defined focal area of the rectum in subjects treated with EPA compared to subjects receiving placebo.
Time Frame: 6 months compared to baseline.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of change in total polyps
Groups:
- 2g/Day Eicosapentanoic Acid (EPA): Eicosapentanoic Acid (EPA): 2 x 500mg EPA capsules twice daily for 6 months
  Endoscopy: With video and photographs at baseline and month 6.
  Biopsies taken: 9 biopsies taken at baseline and month 6 from the rectum of normal mucosa for analysis of apoptosis (3 biopsies), cell proliferation (3 biopsies) and mucosal fatty acid levels (3 biopsies). Two biopsies taken at baseline and month 6 from polyps for cell proliferation (1 biopsy) and apoptosis (1 biopsy).
Arm/Group | 2g/Day Eicosapentanoic Acid (EPA) | Placebo
Number analyzed (Participants) | 23 | 22
percentage of change in total polyps | -12.6 [-24.7 to -0.6] | 9.7 [-2.6 to 22.0]

3. Secondary Outcome: Change in Global Rectal Polyp Burden.
Description: Change in global rectal polyp burden in subjects treated with Eicosapentanoic Acid (EPA) compared to subjects receiving placebo. Each reviewer in the Polyp Video Scoring Committee assessed global colorectal polyp burden change as "better", "same as" or "worse". The qualitative assessment was assigned a score of +1 for "better", 0 for "same as" and -1 for "worse". Thereafter a mean overall reviewers score was calculated.
Time Frame: 6 months compared to baseline.
Population: 5 subjects in the full analysis set lacked the video required for determining global rectal polyp burden due to failure of equipment.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 2g/Day Eicosapentanoic Acid (EPA) | Placebo
Number analyzed (Participants) | 25 | 25
units on a scale | 0.09 [-0.14 to 0.32] | -0.34 [-0.56 to -0.11]

4. Secondary Outcome: Relative EPA Concentration of Total Free Fatty Acids in the Rectal Mucosa.
Description: Relative EPA concentration of total free fatty acids in the rectal mucosa of subjects with FAP.
Time Frame: 6 months compared to baseline.
Population: 3 subjects in the full analysis set had no samples for analysis.
Measure: Mean (95% Confidence Interval); unit: percentage of total fatty acid content
Arm/Group | 2g/Day Eicosapentanoic Acid (EPA) | Placebo
Number analyzed (Participants) | 26 | 26
percentage of total fatty acid content | 1.56 [0.97 to 2.15] | 0.54 [-0.06 to 1.13]

5. Secondary Outcome: Number of Subjects With Adverse Events.
Description: Incidence of adverse events in each treatment group.
Time Frame: 6 months compared to baseline
Measure: Number; unit: participants
Arm/Group | 2g/Day Eicosapentanoic Acid (EPA) | Placebo
Number analyzed (Participants) | 29 | 29
participants | 25 | 25

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | 2g/Day Eicosapentanoic Acid (EPA) | Placebo
Serious Adverse Events (participants affected / at risk) | 3/29 | 0/29
Other Adverse Events (participants affected / at risk) | 25/29 | 25/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2g/Day Eicosapentanoic Acid (EPA) (N=29) | Placebo (N=29)
Small bowel obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0) — Acute small bowel obstruction associated with underlying disease.
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Not related to study medication.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2g/Day Eicosapentanoic Acid (EPA) (N=29) | Placebo (N=29)
Eye disorders (Eye disorders) | 0 (0) | 1 (1) — Episcleritis
Endocrine disorders (Endocrine disorders) | 1 (1) | 0 (0) — Hypothyroidism.
Gastrointestinal (Gastrointestinal disorders) | 23 (68) | 22 (61) — Most common: Abdominal distension. Abdominal pain. Abdominal pain upper. Diarrhoea. Dyspepsia. Faeces discoloured. Flatulence. Nausea. Stomach discomfort. Vomiting.
General disorders (General disorders) | 7 (8) | 9 (11) — Chills. Fatigue. Hemia. Influenza-like illness. Malaise. Pain. Thirst.
Immune system disorders (Immune system disorders) | 1 (1) | 0 (0) — Seasonal allergy
Infections and infestations (Infections and infestations) | 8 (11) | 7 (7) — Ear infection. Gastroenteritis viral. Infected cyst. Infection localised. Influenza. Localised infection. Lower respiratory tract infection. Naso-pharyngitis. Skin infection. Tonsillitis. Tooth abscess. Tracheitis. Baricella
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) — Back injury. Foot fracture. Neck injury. Procedural pain. Whip lash injury.
Investigations (Investigations) | 1 (1) | 5 (5) — Blood cholesterol increase. Blood creatinine increase. Blood potassium decreased. Lipids increased. Weight decreased. Weight increased.
metabolism and nutritional disorders (Metabolism and nutrition disorders) | 1 (1) | 2 (2) — Decreased appetite.
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 7 (10) | 8 (9) — Arthralgia. Axillary mass. Back pain. Bone cyst. Groin pain. Limb discomfort. Muscle spasms. Musculoskeletal pain. Myalgia. Neck pain. Pain in extremity. Pain in jaw.
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) — Breast cancer. Osteoma.
Nervous system disorders (Nervous system disorders) | 11 (19) | 6 (6) — Dizziness. Dysgeusia. Headache. Migraine
Psychiatric disorders (Psychiatric disorders) | 0 (0) | 2 (2) — Anxiety. Mood swings.
Renal and urinary disorders (Renal and urinary disorders) | 1 (1) | 0 (0) — Pollakiuria.
Reproductive system and breast disorders (Reproductive system and breast disorders) | 0 (0) | 3 (3) — Breast mass. Epididymal cyst. Mensturation irregular.
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4) — Cough. Epistaxis. Increased upper airways secretion. Pharyngolaryngeal pain.
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) — Heal rash. Rash.
Vascular disorders (Vascular disorders) | 0 (0) | 1 (1) — Hot flush.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less